CLINICAL TRIAL: NCT00666627
Title: A 2-year Randomised Parallel Group Trial of Alendronate, Ibandronate and Risedronate for Postmenopausal Osteoporosis in Secondary Care.
Brief Title: Bisphosphonate Action on the Appendicular Skeleton: Evidence for Differential Effects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Procter and Gamble (Industry); University of Sheffield (Other)
Responsible Party: Professor Richard Eastell, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH 14463
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Post-menopausal Osteoporosis
Keywords: Osteoporosis; Post-menopausal osteoporosis; Bisphosphonates; Alendronate; Ibandronate; Risedronate
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Ibandronic Acid; Risedronic Acid; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Ibandronate
  Interventions: Drug: Ibandronate
- 2 (Active Comparator): Risedronate
  Interventions: Drug: Risedronate
- 3 (Active Comparator): Alendronate 70mg once weekly
  Interventions: Drug: Alendronate
- 4 (No Intervention): Young women control group

INTERVENTIONS:
Drug: Ibandronate — once monthly
  Other Names: Bonviva
  Arms: 1
Drug: Risedronate — Risedronate 35mg once weekly
  Other Names: Actonel
  Arms: 2
Drug: Alendronate — Alendronate 70mg once weekly
  Other Names: Fosamax
  Arms: 3

SUMMARY:
A study to determine if the three licensed bisphosphonates (alendronate, ibandronate and risedronate):a) affect the peripheral skeleton differently, as assessed by quantitative ultrasound of bone (QUS), peripheral quantitative computed tomography (pQCT) and dual-energy x-ray absorptiometry (DXA)? b) have different effects on bone cells and their activity as assessed by flow cytometry and biochemical markers of bone cell activity? The aim of the study is to compare the effects of three licensed bisphosphonates on bone quantity and quality. There has been no such study before. Most of the measures of bone quantity and quality used in this protocol have not been studied with any of these three agents. The novelty of the study necessitates the establishment of reference ranges and this explains the need for the inclusion of a group of young women.

DETAILED DESCRIPTION:
There have been a number of randomised controlled trials examining the effect of bisphosphonates on fracture risk. The results of these trials have not been uniform, especially in relation to non-vertebral fractures. We have proposed that much of the fracture risk reduction with risedronate can be explained by the reduction in bone resorption markers (Eastell et al, 2003). Each of these three bisphosphonates reduces bone resorption markers, and alendronate and ibandronate are at least as effective as risedronate in this regard. However, there have been few direct comparisons of the different bisphosphonates on surrogate endpoints such as bone mineral density and bone turnover markers. This raises the question of whether the bisphosphonates might affect some other aspect of bone strength, such as 'bone quality'.

The purpose the study is to determine whether three licensed bisphosphonates affect the skeleton differently using a variety of methods (various bone densitometry devices and ultrasound measurements of the bone) at a variety of bone sites (spine, hip, fingers, heel, forearm and leg). These changes will be compared to changes in other markers of bone health such as biochemical markers of bone turnover to help us determine the possible mechanism of action for the different treatments. The study will last for 48 weeks which should be long enough to detect signfiicant changes on bone strength as measured by DXA at the spine/hip. As we are interested in how these changes occur there are more visits in the first three months of the study than the last 9 months of the study. This is expected to help us detect the difference between the onset of the effects of the three treatments more clearly.

Study vists will be: screening, baseline 1, baseline 2, 1 week, 2 weeks, 4 weeks, 12 weeks, 13 weeks (phone calls to participants at 24 and 36 weeks), 48 weeks and 49 weeks. The two baseline visits will allow duplicate measurements of bone stregth/quality on different occasions at the start of the study to minimise variability. Treatment will begin at baseline 2 (0 days) and last for 48 weeks. The visits at 13 weeks and 49 weeks are to perform bone density/quality tests in duplicate to minimise variability as at baseline visit.

Bone mineral density of various bones (hip/spine/whole body and forearm) will be measured by DXA on various devices, quantitative ultrasound will be performed at the heel and fingers, and bone quality will be measured by pQCT at the forearm and tibia/3D analysis of the hip scans at the baseline visits, at 12 and 13 weeks and at 48 and 49 week visits Surrogate markers of bone health (biochemical markers of bone turnover) will be measured at baseline, 1, 2 4, 12, 13, 48 and 49 weeks. Exploratory methods included in the protocol include: Assessing the number of bone breaking down cell numbers (osteoclasts) at baseline, 1 week and 48 weeks Assessing nail brittleness at baseline 12 and 48 weeks.

Subjects will be randomised using a stratification method to ensure all groups have an equal range of bone strength at study entry. Randomisation will be performed by the hospital pharmacy. The study is not blinded and subjects will know which treatment they are on. Subjects will be asked not to discuss their assigned treatment with staff performing bone measurements. There is no placebo group in this trial as all subjects will taking one of the three treatments. We have chosen the active comparator design as many of the measurements (especially the biochemical and cellular ones) do not change unless treatment is given; also, these treatments are indicated and effective in this patients group.

To generate control data we will recruit a group of 200 healthy young women aged 35-40 years. The control group will undertake all the measurements of bone strength/quality that the treatment group will have as well as the biochemical maerkers of bone turnover. There will be only 2 study visits for the control group,baseline and 48 weeks. This data will serve as internal controls and as reference ranges for each of the devices used in the study. Ethical considerations for this study include the use of ionising radiation, blood sampling at each study visit and the number of study visits. This may be balanced by the close monitoring of the subject whilst on the study and a thorough assessment of bone health for 49 weeks. Research participants, patient groups or communities were not involved in the design of this research study.

The hypothesis of the study is that bisphosphonates have varying magnitude of effect on non-vertebral fractures and this is reflected in different changes in measures of bone quality (QUS), bone density in the appendicular skeleton (DXA and pQCT) and novel biochemical markers of bone resorption and osteoclast precursors.

ELIGIBILITY:
Inclusion Criteria:

* be female
* at least 5 years post menopausal but <85 years
* BMD T-score (at the lumbar spine or total hip) of less than or equal to

  * 2.5, or T-score less than or equal to -1 with a low trauma fracture.
* be ambulatory
* be able and willing to participate in the study and provide written informed consent

Exclusion Criteria:

* have evidence of a clinically significant organic disease which could prevent the patient from completing the study
* have a BMI less than 18 or greater than 35
* abuse alcohol or use illicit drugs or who consumed more than 4 servings of any alcoholic beverage one day prior to the visit (i.e., subjects who might be binge drinkers)
* have any history of cancer within the past 5 years excluding skin cancer non melanomas
* have a history of ongoing conditions or diseases known to cause abnormalities of calcium metabolism or skeletal health (secondary osteoporosis)
* Chronic renal disease (as defined by a creatinine clearance of ≤ 30ml/min)
* Acute or chronic hepatic disease
* Malabsorption syndromes
* Hyperthyroidism as manifested by TSH outside the lower limit of the normal range
* Hyperparathyroidism
* Hypocalcemia or hypercalcemia
* Osteomalacia
* Cushing's syndrome
* Patient who are currently on glucocorticoid therapy
* have a serum calcium less than 2.2 mmol/l and a PTH above 75ng/l
* have a history of any known condition that would interfere with the assessment of DXA at either lumbar spine or femoral neck
* have markedly abnormal clinical laboratory parameters that are assessed as clinically significant by the investigator
* use any of the following medications within 12 months of starting study drug

  * Bisphosphonates (at any dose)
  * Use of any fluoride with the exception use for oral hygiene
  * Strontium
  * Other bone agents (i.e., SERM, isoflavones, HRT etc)
* have participated in another clinical trial involving active therapy 3 months prior to randomisation
* have a history of allergic reaction to bisphosphonates
* patient taking calcium supplements within the last month prior to randomisation
* We will exclude patients with secondary osteoporosis, those who have been on anti-resorptive treatments in the past year, and women less than 5 years since menopause, and those with bilateral fractures in the measurement regions (heel, hip and forearm).
* Have suffered a recent fracture within the last 12 months

Ages: 35 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2007-04 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in heel broadband ultrasound attenuation | 2 years

SECONDARY OUTCOMES:
Changes in the percentage of MCSFR+ monocytes in the peripheral blood at baseline and after one week and 48 weeks of therapy | 2 years
Change in SOS at finger and heel at 48 weeks. | 2 years
Change in lumbar spine and total hip BMD measured by DXA at 48 weeks | 2 years
Change in finger BMD measured by RA at 48 weeks | 2 years
Change in heel BMD measured by DXL at 48 weeks | 2 years
Change in distal tibia and ultradistal forearm cortical and trabecular volumetric BMD by pQCT at 48 weeks | 2 years
Changes in cathepsin K and MM enzyme and OPG and RANK-L protein at 12 weeks | 12 weeks
Changes in uNTX and uCTX. At 12 weeks | 12 weeks
Change in disulfide bond content of nails at 48 weeks | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eugene McCloskey, Dr, Study Director — University of Sheffield; Rosemary Hannon, Dr, Study Director — University of Sheffield; Angela Rogers, Dr, Study Director — University of Sheffield; Margaret Paggiosi, Dr, Study Director — University of Sheffield
Locations (1):
- Academic Unit of Bone Metabolism (Sheffield), Sheffield, South Yorkshire, United Kingdom